CLINICAL TRIAL: NCT02970760
Title: Computer Assisted Measurement of Colorectal Polyps
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: CAMP
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colonic polyps
Oversight: Data Monitoring Committee: No

SUMMARY:
Adenomas are polyps of the colorectum that have the potential to develop into colon cancer. However, some adenomas never become malignant tumors, or if so, progression from adenoma into cancer takes a long time. As a result, screening colonoscopy programs were established in order to detect and resect adenomas at an early stage. After resection, polyps should be sent to pathology in order to make a histological diagnosis. Approximately 40-50% of all polyps have adenomatous histology whereas others contain benign histology (e.g. hyperplastic or inflammatory polyps). The latter polyps do not bear the risk to develop colon cancer.

The bigger a polyp is the greater the chance is of it being malignant. During colonoscopy polyp size can be estimated visually by comparing the polyp with an opened biopsy forceps. The span of an opened forceps is 7 mm. Prior to using this technique, the forceps has to be inserted into the colon through a small working channel of the endoscope. Information on the actual adenoma size is crucial as surveillance recommendations depend on the size of the resected polyps. Moreover current guidelines contain the possibilities to disregard hyperplastic polyps in the sigmoid colon if the polyp size is below 5 mm. This means that diminutive hyperplastic polyps (< 5mm) do not necessarily require resection due to their benign dignity. However, there is increasing evidence that large human bias effects exist in estimating the size of polypoid lesions. For example, it has been shown that endoscopists exhibit terminal digit preferences leading to an exaggeration of estimated polyp size. In consequence the human bias problem might lead to wrong adenoma surveillance decisions.

There is no doubt that technical devices are needed which can support endoscopists in finding the right declaration of polyp sizes. The aim of the current project is to create a computer program that is able to automatically measure polyp sizes during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy
* patients >= 18 years

Exclusion Criteria:

* pregnant women
* indication for colonoscopy: inflammatory bowel disease
* indication for colonoscopy: polyposis syndrome
* indication for colonoscopy: emergency colonoscopy e.g. acute bleeding
* contraindication for polyp resection e.g. patients on warfarin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Polyp size as assessed by the computer program | up to 2 weeks
  The predicted polyp size (made by the computer program) will be assessed; the size will be compared with the actual polyp size (as assessed by endoscopist = gold standard). Participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No